CLINICAL TRIAL: NCT01557920
Title: The Effects of Sevoflurane, Propofol, and Carbon Dioxide 'Reversal' on Upper Airway Collapsibility in Healthy, Adult Subjects
Brief Title: The Effects of General Anesthetics on Upper Airway Collapsibility in Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Matthias Eikermann, Director of Research, Surgical Intensive Care Unit, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2011P002472
Record Dates: First submitted 2012-03-15; First posted 2012-03-20 (Estimated); Results first posted 2016-04-21 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-08

CONDITIONS: Airway Complication of Anaesthesia; Healthy
Keywords: apnea; airway collapsibility; healthy; hypercapnia; general anesthesia; breathing-swallow coordination; aspiration
MeSH Terms: conditions — Apnea; Hypercapnia | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol (Active Comparator): The healthy subject will be anesthetized with Propofol. Respiratory measurements will be taken while the subject is anesthetized to calculate the airway closing pressure. After recovery from anesthesia, airway diameter and duty cycle will also be measured. In addition to breathing air mixture, subject will be given carbon dioxide to achieve end tidal CO2 levels of 4 mm and 8 mm above baseline. All respiratory measurements will be repeated at each level above baseline. Assessment of swallow patterns during anesthesia and wakefulness, as well as under differential CO2 levels will be assessed offline after recovery from anesthesia.
  Interventions: Drug: Propofol
- Sevoflurane (Active Comparator): The healthy subject will be anesthetized with Sevoflurane. Respiratory measurements will be taken while the subject is anesthetized to calculate the airway closing pressure. After recovery from anesthesia, airway diameter and duty cycle will also be measured. In addition to breathing air mixture, subject will be given carbon dioxide to achieve end tidal CO2 levels of 4 mm and 8 mm above baseline. All respiratory measurements will be repeated at each level above baseline. Assessment of swallow patterns during anesthesia and wakefulness, as well as under differential CO2 levels will be assessed offline after recovery from anesthesia.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — Propofol administration for induction of general anesthesia. Administration will be performed IV, using a Target Controlled Induction Pump.
  Arms: Propofol
Drug: Sevoflurane — Sevoflurane will be administered via mask inhalation to achieve anesthesia.
  Arms: Sevoflurane

SUMMARY:
The investigators hypothesize that propofol, when compared to sevoflurane, causes the upper airway to collapse more easily and causes less activity in the tongue muscle. Additionally, the investigators hypothesize that, under increased carbon dioxide concentrations of the air inhaled, the upper airway will be less likely to collapse under anesthesia and there will be increased activity in the tongue muscle under both propofol and sevoflurane, when compared to breathing normal concentrations of carbon dioxide, as in room air. Furthermore the investigators hypothesize that anesthesia disrupt the breathing swallow coordination, an effect additionally altered by increased carbon dioxide through increased respiratory drive.

DETAILED DESCRIPTION:
Upper airway patency depends on an appropriate balance between the dilating force of pharyngeal muscles and the collapsing force of negative intraluminal pressure, which is generated by respiratory "pump" muscles. The genioglossus (GG) protects pharyngeal patency in humans. This muscle receives various types of neural drive, distributed differentially across the hypoglossal motoneuron pool, including phasic (inspiratory) and tonic (non-respiratory) drives. In addition, reflex GG activation in response to negative pharyngeal pressure stabilizes upper airway patency both in humans and in rats. General anesthetic agents, including propofol and sevoflurane, predispose the upper airway to collapse, at least in part by decreasing upper airway muscle activity.

Theoretically anesthetics could affect upper airway dilator activity by several mechanisms, including an anesthetic-induced, dose-dependent decrease in hypercapnic and hypoxic ventilatory drive, hypoglossal motoneuron depression, decreased skeletal muscle contractility, an increase in phasic GG activity as a result of decreased arterial blood pressure, and an increase in phasic hypoglossal nerve discharge.

Previous studies have shown that certain anesthetics, including pentobarbital and isoflurane, can increase genioglossus phasic activity in rats and in humans. The effects of propofol on airway collapsibility have been studied in humans however, to our knowledge, they have not been measured under conditions of hypercapnia. Studies of airway collapsibility under sevoflurane anesthesia have been performed in children, but no data exists for airway collapsibility in sevoflurane-anesthetized adults. Similarly no data exists on the effects of sevoflurane on GG activity

In a previous trial of pentobarbital-anesthetized volunteers, the investigators observed that mild hypercapnia (5 - 10 mmHg above baseline) produced a significant increase in flow rate and GG phasic activity, as well as a smaller increase in GG tonic activity. If our proposed study shows a beneficial effect, then the investigators plan a follow-up study addressing the possibility that hypercapnia may be used therapeutically for airway protection. A similar concept has already been considered for critically ill ICU patients.

However, previous studies have shown that a hypercapnia-induced increase in ventilatory drive can inhibit airway protective reflexes by disrupting the breathing swallowing coordination. In order to assess the safety of induced mild hypercapnia as an intervention for airway protection, we evaluated whether variable levels of hypercapnia occurring during anesthesia with sevoflurane and propofol impair the coordination of breathing and swallowing compared with the effects of anesthesia alone.

With this pharmaco-physiological interaction study on healthy adults we aim to:

1. Compare the effects of sevoflurane and propofol on upper airway closing pressure, upper airway muscle control and breathing.
2. Assess the effects of evoked hypercapnia (carbon dioxide reversal) on propofol-induced upper airway collapsibility
3. Evaluate the effects of sevoflurane, propofol, and induced hypercapnia on coordination of breathing and swallowing.

Comparative drug studies on airway effects of anesthetics in humans are important for defining an optimal anesthetic regimen for patients at risk of airway collapse, such as patients with obstructive sleep apnea. Our studies are also particularly relevant for patients undergoing procedural sedation, which is typically being conducted under spontaneous ventilation with the upper airway being unprotected. In addition, our results may increase our understanding of postoperative airway obstruction, a common complication in the post-anesthesia recovery room.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class I
* Age between 18 and 45
* BMI 18-28 kg/m^2

Exclusion Criteria:

* Concurrent significant medical illness (heart disease including untreated hypertension, Clinically significant kidney disease, liver disease, or lung disease, History of myasthenia gravis or other muscle and nerve disease)
* Anxiety disorder requiring treatment
* Concurrent medications known to affect anesthesia, upper airway muscles or respiratory function (e.g., gabaergic anxiolytics, antipsychotics)
* Individuals with a history of allergy or adverse reaction to lidocaine, propofol, or sevoflurane
* For women: pregnancy
* Suggestion of obstructive sleep apnea (OSA) or any other sleep disorder (e.g. witnessed apneas, gasping or choking during sleep, unexplained excessive daytime sleepiness)
* History of drug or alcohol abuse
* Acute intermittent porphyria

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-01; Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Eikermann, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Eikermann M, Malhotra A, Fassbender P, Zaremba S, Jordan AS, Gautam S, White DP, Chamberlin NL. Differential effects of isoflurane and propofol on upper airway dilator muscle activity and breathing. Anesthesiology. 2008 May;108(5):897-906. doi: 10.1097/ALN.0b013e31816c8a60. PMID 18431126
- [Background] Eikermann M, Grosse-Sundrup M, Zaremba S, Henry ME, Bittner EA, Hoffmann U, Chamberlin NL. Ketamine activates breathing and abolishes the coupling between loss of consciousness and upper airway dilator muscle dysfunction. Anesthesiology. 2012 Jan;116(1):35-46. doi: 10.1097/ALN.0b013e31823d010a. PMID 22108392
- [Background] Eikermann M, Eckert DJ, Chamberlin NL, Jordan AS, Zaremba S, Smith S, Rosow C, Malhotra A. Effects of pentobarbital on upper airway patency during sleep. Eur Respir J. 2010 Sep;36(3):569-76. doi: 10.1183/09031936.00153809. Epub 2009 Dec 23. PMID 20032012

RESULTS

PARTICIPANT FLOW:
Groups:
- Propofol First, Then Sevoflurane: The healthy subject will be anesthetized first with Propofol, and secondarily with Sevoflurane. Respiratory measurements will be taken while the subject is anesthetized to calculate the airway closing pressure. After recovery from anesthesia, airway diameter and duty cycle will also be measured. In addition to breathing air mixture, subject will be given carbon dioxide to achieve end tidal CO2 levels of 4 mm and 8 mm above baseline. All respiratory measurements will be repeated at each level above baseline.
  Propofol: Propofol administration for induction of general anesthesia. Administration will be performed IV, using a Target Controlled Induction Pump.
  Sevoflurane: Sevoflurane will be administered via mask inhalation to achieve anesthesia.
- Sevoflurane First, Then Propofol: The healthy subject will be anesthetized first with Sevoflurane, and secondarily with Propofol. Respiratory measurements will be taken while the subject is anesthetized to calculate the airway closing pressure. After recovery from anesthesia, airway diameter and duty cycle will also be measured. In addition to breathing air mixture, subject will be given carbon dioxide to achieve end tidal CO2 levels of 4 mm and 8 mm above baseline. All respiratory measurements will be repeated at each level above baseline.
  Propofol: Propofol administration for induction of general anesthesia. Administration will be performed IV, using a Target Controlled Induction Pump.
  Sevoflurane: Sevoflurane will be administered via mask inhalation to achieve anesthesia.
Period: Overall Study
Arm/Group | Propofol First, Then Sevoflurane | Sevoflurane First, Then Propofol
Started | 9 | 9
Completed | 6 | 6
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Crossover Randomized Propofol and Sevoflurane: The healthy subject will be anesthetized with Propofol and Sevoflurane in a randomized crossover fashion. Respiratory measurements will be taken while the subject is anesthetized to calculate the airway closing pressure. After recovery from anesthesia, airway diameter and duty cycle will also be measured. In addition to breathing air mixture, subject will be given carbon dioxide to achieve end tidal CO2 levels of 4 mm and 8 mm above baseline. All respiratory measurements will be repeated at each level above baseline.
  Spontaneous swallows were identified, and categorized as physiological or pathological. Physiological swallows were followed by expiratory flow (E or I-E). Pathological swallows were followed by inspiration (I and E-I).
  Propofol: Propofol administration for induction of general anesthesia. Administration will be performed IV, using a Target Controlled Induction Pump.
  Sevoflurane: Sevoflurane will be administered via mask inhalation to achieve anesthesia.
Arm/Group | Crossover Randomized Propofol and Sevoflurane
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Upper Airway Closing Pressure
Description: Upper airway closing pressure will be measured during steady state anesthesia as well as during carbon dioxide reversal.
Time Frame: participants will be followed for the duration of anesthesia, an expected average of 6 hours
Population: Ten out of 12 subjects were analyzed. In two subjects we could not record high quality biologically plausible recordings of upper airway closing pressure. Data from multiple measurements per participant were combined to calculate an average upper airway closing pressure per subject.
Measure: Mean (Standard Deviation); unit: cm H20
Groups:
- Propofol: The healthy subject will be anesthetized with Propofol. Respiratory measurements will be taken while the subject is anesthetized to calculate the airway closing pressure. After recovery from anesthesia, airway diameter and duty cycle will also be measured. In addition to breathing air mixture, subject will be given carbon dioxide to achieve end tidal CO2 levels of 4 mm and 8 mm above baseline. All respiratory measurements will be repeated at each level above baseline.
  Propofol: Propofol administration for induction of general anesthesia. Administration will be performed IV, using a Target Controlled Induction Pump.
- Sevoflurane: The healthy subject will be anesthetized with Sevoflurane. Respiratory measurements will be taken while the subject is anesthetized to calculate the airway closing pressure. After recovery from anesthesia, airway diameter and duty cycle will also be measured. In addition to breathing air mixture, subject will be given carbon dioxide to achieve end tidal CO2 levels of 4 mm and 8 mm above baseline. All respiratory measurements will be repeated at each level above baseline.
  Sevoflurane: Sevoflurane will be administered via mask inhalation to achieve anesthesia.
Arm/Group | Propofol | Sevoflurane
Number analyzed (Participants) | 10 | 10
cm H20 | -9.83 (3.92) | -10.77 (4.69)

2. Primary Outcome: Proportion of Pathological Swallows
Description: A pathological swallow was defined as a swallow that was followed by inspiratory flow. A physiological swallow was defined as a swallow that was followed by expiratory flow. The number of pathological and physiological swallows were measured during wakefulness and anesthesia. The pathological swallows are presented as percentage of path. swallows calculated as path.sw/[path.sw+phys.sw]*100 (%).
Time Frame: swallows were measured during steady state conditions (mean±SEM, 2.6±0.6h)
Population: 224 swallows in 11 out of 12 subjects were analyzed (1 excluded due to faulty recording of swallows).
Measure: Number; unit: percentage of pathological swallows
Groups:
- Anesthesia With Propofol and Sevoflurane (All Cases): Proportion of pathological (inspiratory) swallows during anesthesia with propofol and sevoflurane (across carbon-dioxide (CO2) levels).
- Wakefulness (All Cases): Proportion of pathological (inspiratory) swallows during wakefulness (across CO2 levels)
- Anesthesia With Propofol and Sevoflurane (Baseline CO2): Proportion of pathological (inspiratory) swallows during anesthesia with propofol and sevoflurane (during baseline CO2).
- Anesthesia With Propofol and Sevoflurane (CO2 Insufflation): Proportion of pathological (inspiratory) swallows during anesthesia (with CO2+4 and +8 insufflation).
- Wakefulness (During Baseline CO2): Proportion of pathological (inspiratory) swallows during anesthesia (during baseline CO2).
- Wakefulness (With CO2 Insufflation): Proportion of pathological (inspiratory) swallows during wakefulness (with CO2+4 and +8 insufflation).
Arm/Group | Anesthesia With Propofol and Sevoflurane (All Cases) | Wakefulness (All Cases) | Anesthesia With Propofol and Sevoflurane (Baseline CO2) | Anesthesia With Propofol and Sevoflurane (CO2 Insufflation) | Wakefulness (During Baseline CO2) | Wakefulness (With CO2 Insufflation)
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 11 | 11
percentage of pathological swallows | 25.9 | 4.9 | 15.8 | 34.9 | 1.0 | 13.2
Statistical Analysis 1: Comparison: Anesthesia With Propofol and Sevoflurane (All Cases) vs Wakefulness (All Cases); Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — pathological swallows under anesthesia vs. wakefulness: 25.9% vs. 4.9%
Statistical Analysis 2: Comparison: Anesthesia With Propofol and Sevoflurane (Baseline CO2) vs Anesthesia With Propofol and Sevoflurane (CO2 Insufflation) vs Wakefulness (During Baseline CO2) vs Wakefulness (With CO2 Insufflation); Comparison of pathological swallow-rate increase by carbon-dioxide during anesthesia and wakefulness; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

3. Secondary Outcome: Airway Diameter
Description: Using acoustic pharyngometry, we intend to measure the cross-sectional area of the airway at several points during recovery from anesthesia.
Time Frame: participants will be followed for the duration of anesthesia until full recovery, an expected average of 9 hours
Population: No data were obtained.
Arm/Group | Wakefulness | Anesthesia With Low Dose Sevoflurane (Baseline CO2) | Anesthesia With High Dose Sevoflurane (Baseline CO2) | Anesthesia With Low Dose Propofol (CO2 Baseline) | Anesthesia With High Dose Propofol (CO2 Baseline)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Genioglossus Muscle Electromyogram
Description: will be measured during steady state anesthesia as well as during carbon dioxide reversal, and during recovery from anesthesia.
Time Frame: participants will be followed for the duration of anesthesia until full recovery, an expected average of 9 hours
Population: The number of participants in this group are only 9 since the genioglossus EMG signals were poor in 2 participants and these were excluded from the analysis.
Measure: Mean (Standard Error); unit: percentage of maximum recorded activity
Groups:
- Phasic Genioglossus Activity (Light Anesthesia); Phasic Genioglossus Activity (Deep Anesthesia): Phasic activity (Peak activity - Tonic activity)
- Tonic Genioglossus Activity (Light Anesthesia): Tonic Genioglossus activity (light anesthesia)
- Tonic Genioglossus Activity (Deep Anesthesia): Tonic Genioglossus activity (deep anesthesia)
Arm/Group | Phasic Genioglossus Activity (Light Anesthesia) | Tonic Genioglossus Activity (Light Anesthesia) | Phasic Genioglossus Activity (Deep Anesthesia) | Tonic Genioglossus Activity (Deep Anesthesia)
Number analyzed (Participants) | 9 | 9 | 9 | 9
percentage of maximum recorded activity | 32.8 (2.1) | 24.2 (1.8) | 26.0 (1.8) | 22.3 (2.0)

5. Secondary Outcome: Minute Ventilation (Tidal Volume and Respiratory Rate)
Description: Measured by spirometry. Subjects wear a full-face mask. Reported in L/min
Time Frame: Will be measured before and during anesthesia until emergence from anesthesia, an expected average of 6 hours
Population: In one subject we could not record high quality biologically plausible recordings of minute ventilation.
Measure: Mean (Standard Deviation); unit: L/min
Groups:
- Wakefulness: Minute Ventilation (CO2 baseline)
- Anesthesia With Low Dose Sevoflurane (Baseline CO2): Minute ventilation during anesthesia with sevoflurane (during baseline CO2).
- Anesthesia With High Dose Sevoflurane (Baseline CO2): Minute ventilation during anesthesia with sevoflurane (baseline CO2)
- Anesthesia With Low Dose Propofol (CO2 Baseline): Minute Ventilation during anesthesia with propofol (CO2 baseline).
- Anesthesia With High Dose Propofol (CO2 Baseline): Minute Ventilation during anesthesia with propofol (during baseline CO2).
Arm/Group | Wakefulness | Anesthesia With Low Dose Sevoflurane (Baseline CO2) | Anesthesia With High Dose Sevoflurane (Baseline CO2) | Anesthesia With Low Dose Propofol (CO2 Baseline) | Anesthesia With High Dose Propofol (CO2 Baseline)
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 11
L/min | 7.9 (1.7) | 6.7 (1.3) | 5.6 (1.5) | 7.2 (1.7) | 5.7 (1.3)

6. Secondary Outcome: Duty Cycle
Description: (T(ins)/T(total))*100
Time Frame: Will be measured before and during anesthesia until emergence from anesthesia, an expected average of 6 hours
Population: In one subject we could not record high quality biologically plausible recordings of Duty cycle.
Measure: Mean (Standard Deviation); unit: percentage of Ttotal
Groups:
- Wakefulness: Duty cycle (CO2 baseline)
- Anesthesia With Low Dose Sevoflurane (Baseline CO2): Duty cycle during anesthesia with sevoflurane (during baseline CO2).
- Anesthesia With High Dose Sevoflurane (Baseline CO2): Duty cycle during anesthesia with sevoflurane (baseline CO2)
- Anesthesia With Low Dose Propofol (CO2 Baseline): Duty cycle during anesthesia with propofol (CO2 baseline).
- Anesthesia With High Dose Propofol (CO2 Baseline): Duty cycle during anesthesia with propofol (during baseline CO2).
Arm/Group | Wakefulness | Anesthesia With Low Dose Sevoflurane (Baseline CO2) | Anesthesia With High Dose Sevoflurane (Baseline CO2) | Anesthesia With Low Dose Propofol (CO2 Baseline) | Anesthesia With High Dose Propofol (CO2 Baseline)
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 11
percentage of Ttotal | 42 (3) | 42 (5) | 43 (4) | 40 (3) | 41 (3)

7. Post Hoc Outcome: Frequency of Spontaneous Swallows During Anesthesia vs Wakefulness
Description: The number of swallows were counted during wakefulness and anesthesia. The frequency of swallowing was calculated per hour
Time Frame: swallows were measured during steady state conditions (mean±SEM, 2.6±0.6h)
Population: 224 swallows in 11 out of 12 subjects were analyzed (1 excluded due to faulty recording of swallows). If the pathological swallow incidence between sevoflurane and propofol anesthesia had a p-value >0.05, subsequent analyses were conducted to evaluate depth of anesthesia related differences rather than compound specific ones.
Measure: Mean (Standard Deviation); unit: number of swallows/hr
Arm/Group | Anesthesia With Propofol and Sevoflurane | Wakefulness
Number analyzed (Participants) | 11 | 11
number of swallows/hr | 1.7 (3.3) | 28 (22.3)
Statistical Analysis 1: Comparison: Anesthesia With Propofol and Sevoflurane vs Wakefulness; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The number of swallows per hour: 1.7±3.3 during anesthesia vs. 28.0±22.3 during wakefulness

ADVERSE EVENTS:
Arm/Group | Propofol | Sevoflurane
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes